CLINICAL TRIAL: NCT06168188
Title: Principle Investigator Initiated Clinical Trial: The Neuroprotective Effect of Novel Long-acting Granulocyte-colony-stimulating Factor (PEG-GCSF) in the Traumatic Optic Neuropathy
Brief Title: The Neuroprotective Effect of PEG-GCSF in the Traumatic Optic Neuropathy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Rong-Kung Tsai, Professor, Buddhist Tzu Chi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCMF-EP 108-01
Record Dates: First submitted 2021-12-02; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Injuries | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neulasta (Experimental): The 0.15 mL of Neulasta will be filled into 1 mL of syringe equipped with 30 gauge beveled needle for intravitreal injection.
  Interventions: Drug: Neulasta® (pegfilgrastim)

INTERVENTIONS:
Drug: Neulasta® (pegfilgrastim) — Intravitreal injection of Neulasta® (pegfilgrastim) after TON

SUMMARY:
The clinical trial will be a phase 1, semi-experimental trial, which will be performed in Hualien Tzu Chi Hospital. Twenty patients will be recruited in this study starting from the 2nd year of the project to the 3rd year of the project and will go through comprehensive eye and systemic examination in the Hualien Tzu Chi Hospital. Indirect TON (ITON) patients are defined as reduced best corrected visual acuity (BCVA), visual field, color vision, and positive relatively afferent pupillary defect (RAPD) with normal fundus and optic nerve examination and no evidence of direct trauma to optic nerve on spiral orbital and optic canal computer tomography (CT) scan. Therefore, all patients will have examinations of BCVA, visual field, color vision, RAPD, FVEP, CT scan, and IOP for defining ITON patients one day before Neulasta injection. Patient also underwent renal function test, liver function test, coagulation test, and complete blood count before the treatment. Patients who meet the enrollment criteria (inclusion and exclusion) will be fully informed of this treatment and then an informed consent will be obtained. After patient enrolment, the patient will be intravitreally administrated by 0.15 mL of Neulasta in the injured eye. Firstly, the injured eye will be treated with iodine solution for disinfection and then will be treated with Alcaine eye drop for topic anesthesia. The 0.15 mL of Neulasta will be filled into 1 mL of syringe equipped with 30 gauge beveled needle for intravitreal injection. During injection of Neulasta solution, the anterior chamber decompression will be performed for IOP balance. The aqueous humor from anterior chamber will be collected for further microarray analysis. After Neulasta treatment, Tobradex eyedrops (Alcon) will be given on the injected eye, four times a day. Patient will be hospitalized for one day to monitor BCVA, IOP, fundus condition, complete blood count, and any adverse event. During 3-month follow-up trial, each patient will be regularly monitored 7 days and 1, 3 months after treatments by determining the BCVA, the RPAD, the color vision, visual field, the latency of P-100 wave in FVEP, and the RNFL thickness, IOP, and complete blood count.

ELIGIBILITY:
Inclusion Criteria:

1. 20-70 years old
2. Having indirect traumatic optic neuropathy, one week to 4 weeks after trauma
3. Normal disc figure and macula appearance
4. Reduced BCVA (Snellen Chart, less than 20/200) or C-24 central visual field loss more than 10 dB (MD<-10 dB)
5. Color vision defect and positive RAPD
6. No evidence of direct trauma to ON on spiral orbital and optic canal computer tomography (CT) scan.
7. Normal IOP (10-21 mm Hg)
8. Normal blood coagulation (prothrombin time: 8~12s; partial thromboplastin time: 23.9 - 35.5 s; international normalized ratio: 0.85~1.15)
9. Adequate hematologic (absolute neutrophil count ≥1.5 × 109/L, hemoglobin ≥9 g/dL, platelets ≥80 × 109/L, and PT/PTT/INR ≤1.0 × upper limit of normal; ULN)
10. Adequate hepatic function (albumin ≥2.8 g/dL, serum bilirubin ≤2.0 mg/dL or ≤2 × ULN, and aspartate aminotransferase and alanine aminotransferase ≤5.0 × ULN)
11. Adequate renal function (Serum BUN: 6-22 mg/dl; serum creatinine: 0.7-1.5 mg/dl for men, 0.5-1.2 mg/dl for women)
12. No other cranial nerve injuries (cranial nerve examination, nerve number: 1, 3-12)

Exclusion Criteria:

1. Having other injuries that effect on visual function
2. Direct optic neuropathy
3. No light perception
4. Pregnant and breast feeding women
5. Having malignancy
6. Sickle-cell disease
7. G-CSF allergic reaction
8. Acute infectious diseases
9. Benign Intracranial hypertension symptoms (1. papilledema in both eyes with no spontaneous venous pulsation 2. Increase of peripapillary nerve fiber layer thickness in OCT imaging)
10. Associated intracranial hemorrhage or severe skull fracture
11. History or evidence of any other clinically condition that, in the opinion of the investigator, would pose a risk to patient's safety or interfere with study procedures, evaluation, or completion:

    1. Diabetic retinopathy, maculopathy
    2. Uncontrolled hypertension
    3. History of stroke and cardiovascular diseases
    4. Glaucoma

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
BCVA | 3 months after treatment
  Best corrected visual acuity
VA | 3 months after treatment
  Visual Field

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taipei, Not US Or Canada, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu PK, Wen YT, Lin W, Kapupara K, Tai M, Tsai RK. Neuroprotective effects of low-dose G-CSF plus meloxicam in a rat model of anterior ischemic optic neuropathy. Sci Rep. 2020 Jun 25;10(1):10351. doi: 10.1038/s41598-020-66977-9. PMID 32587280
- [Background] Wen YT, Huang TL, Huang SP, Chang CH, Tsai RK. Early applications of granulocyte colony-stimulating factor (G-CSF) can stabilize the blood-optic-nerve barrier and ameliorate inflammation in a rat model of anterior ischemic optic neuropathy (rAION). Dis Model Mech. 2016 Oct 1;9(10):1193-1202. doi: 10.1242/dmm.025999. Epub 2016 Aug 18. PMID 27538969
- [Background] Huang SP, Fang KT, Chang CH, Huang TL, Wen YT, Tsai RK. Autocrine protective mechanisms of human granulocyte colony-stimulating factor (G-CSF) on retinal ganglion cells after optic nerve crush. Exp Eye Res. 2016 Feb;143:132-40. doi: 10.1016/j.exer.2015.10.010. Epub 2015 Oct 28. PMID 26518178
- [Background] Tsai RK, Chang CH, Wang HZ. Neuroprotective effects of recombinant human granulocyte colony-stimulating factor (G-CSF) in neurodegeneration after optic nerve crush in rats. Exp Eye Res. 2008 Sep;87(3):242-50. doi: 10.1016/j.exer.2008.06.004. Epub 2008 Jun 17. PMID 18602391